CLINICAL TRIAL: NCT06251388
Title: A Prospective, Single Arm, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of Concurrent Chemoradiotherapy Followed by Cadonilimab（AK104) for Newly Diagnosed Local Advanced Cervical Cancer
Brief Title: A Study of Concurrent Chemoradiotherapy Followed by Cadonilimab（AK104） for Newly Diagnosed Local Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Collaborators: Afﬁliated Hospital of North Sichuan Medical College (Other); The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Rutie Yin, Clinical Professor, West China Second University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCSUH20231212
Record Dates: First submitted 2024-01-26; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): AK104（10.0 mg/kg，intravenous (IV) infusion，Q3W） after CCRT
  Interventions: Drug: AK104

INTERVENTIONS:
Drug: AK104 — AK104（10.0 mg/kg，intravenous (IV) infusion，Q3W）maintained with no more than 1 year.
  Other Names: Cadonilimab Injection

SUMMARY:
This study will evaluate the efficacy and safety of concurrent chemoradiotherapy（CCRT）followed by cadonilimab（AK104) in high risk local advanced cervical cancer.

Participants received CCRT，efficacy evaluation of CCRT was no disease progression who maintained with AK104（10.0 mg/kg，Q3W）until drug exposure over 1 years or disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* female, Age 18 -75 years.
* Predicted survival ≥ 3 month.
* Histologically and/or cytologically confirmed Squamous cell carcinoma, adenocarcinoma, adenosquamous cell carcinoma, FIGO 2018 stage III-IVA.
* Unable to undergo curative surgery，Pior not received systemic therapy before CCRT, Including but not limited to radiotherapy, chemotherapy, immunotherapy, and biological therapy,etc.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Have at least one evaluable lesion (RECIST 1.1 criteria)
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment.
* participants are eligible to participate if they agree to the contraception use as per study protocol.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Has received other antitumor therapy before CCRT.
* Therapeutic evaluation of CCRT was disease progression.
* Previously received immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, and Ox40 . etc.), immune cell therapy. etc. Any tumor immune mechanisms treatment .
* With brain metastases.
* Previously received allogeneic stem cell or parenchymal organ transplantation.
* Previously or currently suffering from congenital or acquired immunodeficiency diseases.
* known or suspected to have a history of allergies to similar drugs, or has a history of hypersensitivity to chimeric or humanized antibodies or fusion proteins, or is allergic to excipients of the study drug.
* Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive, or HIVAb positive.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* Within the 6 months prior to enrollment, has serious cardiovascular events such as pulmonary embolism, acute myocardial infarction, congestive heart failure (New York Heart Association grade III or IV), and ≥ 2 grade ventricular arrhythmias.
* Cerebrovascular accident within 6 months prior to enrollment.
* Active infection requiring systemic treatment.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, non infectious pneumonia , pulmonary fibrosis, acute lung disease, etc.
* Required systemic treatment with glucocorticoid (>10 mg/day of prednisone or equivalent glucocorticoid) or other immunosuppressive agents within 14 days prior to enter the trial.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Baseline up to approximately 24 months.
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate assessed by Investigator | Baseline up to approximately 12 months.
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR per RECIST v1.1.
Disease control rate | Baseline up to approximately 12 months.
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Overall survival | Baseline up to approximately 48 months.
  OS is the time from randomization to death due to any cause
Safety and adverse reactions of Cadonilimab | Baseline up to approximately 48 months.
  According to CTCAE v5.0, any adverse events that occur to all subjects during the study period will be recorded. We recorded the clinical manifestation characteristics, severity, onset time, duration, treatment method and prognosis, and determined the correlation with Cadonilimab.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China